CLINICAL TRIAL: NCT01188434
Title: Integrating Interventions for Maternal Substance Abuse and Child Neglect
Brief Title: Integrating Interventions for Maternal Substance Abuse
Acronym: ITSAN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Social Learning Center (Other)
Responsible Party: Principal Investigator, Lisa Saldana, Research Scientist, Oregon Social Learning Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23DA021603 (NIH)
Record Dates: First submitted 2010-08-23; First posted 2010-08-25 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Substance Abuse; Child Neglect
Keywords: Methamphetamine; Substance Abuse; Child Neglect; Child Welfare; Evidence Based Practice
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated Behavioral Treatment (Experimental): Combined substance abuse, parenting skills, and basic needs intervention
  Interventions: Behavioral: ITSAN
- casework treatment as usual (Active Comparator): services as usual as referred by child welfare
  Interventions: Behavioral: Services as Usual

INTERVENTIONS:
Behavioral: ITSAN — integrated behavioral intervention for substance abuse, parenting skills, and basic needs
  Arms: Integrated Behavioral Treatment
Behavioral: Services as Usual — Services as usual referred by child welfare
  Arms: casework treatment as usual

SUMMARY:
This Research Plan proposes Stage 1 Research integrating evidence based practices to address the needs of mothers referred to child welfare for substance abuse. Mothers with a history of methamphetamine abuse and child neglect will be recruited. Using an intensive community based treatment, mothers will receive substance abuse treatment combined with parenting skills training and psychosocial support for basic needs (e.g., housing, employment). This project will include a feasibility study (n = 5), followed by a small randomized pilot (n = 24) to examine the efficacy of the Integrated Treatment for Substance Abuse and Neglect compared to treatment as usual, with a population of substance abusing neglectful mothers referred through the Department of Child Welfare.

ELIGIBILITY:
Inclusion Criteria:

* Maternal Substance Abuse
* Child Welfare involvement
* Child Neglect
* English Speaking
* Child either remaining in the home or reunification plan in place
* Living in the county

Exclusion Criteria:

* Current involvement in other substance abuse treatment
* Current involvement in other parenting skills training
* parental rights terminated
* active psychosis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-09; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Addiction Severity Index | Baseline, 6 months, 12 months
  self report of all substances used
Service Utilization Survey | monthly
  self report of social, medical, and mental health services received by parent and youth
Parenting Measures | Baseline, 6 months, 12 months
  Assessment battery of parenting beliefs, expectations, and behaviors

SECONDARY OUTCOMES:
Urinalysis | monthly
  10 panel Urine Drug Screen Collection
Archival data from the Child Welfare system | annually
  System level data of new reports to the child welfare system

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Saldana, PhD, Principal Investigator — OSLC Community Programs
Locations (1):
- OSLC, Eugene, Oregon, United States